CLINICAL TRIAL: NCT00464893
Title: Multicenter, Open-label Phase II Study to Evaluate the Safety and Efficacy of the Trifunctional Bispecific Antibody Catumaxomab (Anti-EpCAM x Anti-CD3) in Patients With Gastric Adenocarcinoma After Neoadjuvant Chemotherapy and Intended Curative Resection
Brief Title: Phase II Study With Catumaxomab in Patients With Gastric Cancer After Neoadjuvant CTx and Curative Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-CAT-GC-03; EudraCT-Nr.:2006-002727-16
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma
Keywords: gastric cancer; catumaxomab; neoadjuvant chemotherapy; phase II; interoperative; trifunctional antibody
MeSH Terms: conditions — Stomach Neoplasms | interventions — catumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- catumaxomab arm (Active Comparator): Patients will get first the chemotherapeutic regimen (Epirubicin, Cisplatin and Capecitabine or 5-Fluorouracil) consisting of three 21-day cycles, starting on the weeks 1, 4 and 7. Four weeks after CTx the D2 surgery will take place. Treatment with catumaxomab will consist of an initial dose of 10µg given intraoperatively as in intraperitoneal bolus and of four postoperative ascending doses.
  Interventions: Drug: Catumaxomab

INTERVENTIONS:
Drug: Catumaxomab — 10 µg intraoperative and 4 ascending doses (10, 20, 50 and 150 µg) on day 7, 10, 13 and 16
  Other Names: Removab
Drug: catumaxomab — 10 µg intraoperatively and 4 ascending doses: 10, 20, 50 and 150 µg
  Other Names: Removab

SUMMARY:
Primary evaluation of the safety, tolerability and feasibility regarding specific postoperative complications of an adjuvant treatment with catumaxomab administered after curative tumor resection subsequent to a neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
An open-label, multi-center phase II study in surgically resectable patients after neoadjuvant ECX-chemotherapy, with confirmed diagnosis of gastric adenocarcinoma and with a high risk of disseminated tumor cells due to serosal infiltration or positive lymph nodes after curative gastrectomy.

Treatment with catumaxomab will consist of an initial dose of 10 µg given intraoperatively as an intraperitoneal bolus and of four postoperative ascending doses (10-20-50-150 µg)which will be administered as an i.p.-infusion using an installed abdominal i.p.-port on the postoperative days 7, 10, 13 and 16.

Catumaxomab is a trifunctional antibody targeting EpCAM on tumor cells and CD3 on T cells. Trifunctional antibodies represent a new concept for targeted anticancer therapy. This new antibody class has the capability to redirect T cells and accessory cells (e.g. macrophages, dendritic cells [DCs] and natural killer [NK] cells) to the tumor site. According to preclinical data, trifunctional antibodies activate these different immune effector cells, which can trigger a complex anti-tumor immune response.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent
* male or female patient at an age of 18 years or older
* patient has a primary diagnosis of a histologically confirmed gastric adenocarcinoma (including GE junction Siewert-Type 2 or 3)
* TNM-staging at screening of T3/T4, N+/-, M0 or T2, N+, M0
* indication and eligibility for a neoadjuvant chemotherapeutic regimen featuring three cycles of ECX with 21 days per cycle
* intended curative gastrectomy
* Karnofsky index > 70

Exclusion Criteria:

* Exposure to prior cancer therapy or planned adjuvant chemo- or radiotherapy of the current gastric cancer
* prior diagnosis of any malignancy not cured by surgery alone less than 5 years before study entry
* previous use of non-humanized monoclonal mouse or rat antibodies
* treatment with another investigational product during this study or during the last 30 days prior to study start
* presence of distant metastases
* presence of constant immunosuppressive therapy
* history of pancreas resection (also partial) or thoracotomy
* presence of any acute or chronic systemic infection
* patient with a bowel obstruction within the last 30 days
* known contraindications to any of the planned ECX chemotherapeutics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
rate of all specific postoperative complications newly observed during a period of 30 days after surgery in those study patients who received at least the first 3 doses of catumaxomab | 30 days after last catumaxomab administration

SECONDARY OUTCOMES:
frequency, relationship and seriousness of adverse events | 30 days after last catumaxomab administration
surgical resection rate | after surgery
chemotherapeutic response rate | after neoadjuvant CTx
overall survival at 3, 6, 9, 12 and 24 month after EOT, defined as the time from study enrolment until death | 2 years
disease-free survival at 3, 6, 9, 12 18 and 24 months after EOT, defined as the time from study enrolment to the point of diagnosis of recurrent disease or death, whichever occurred first | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Bokemeyer, Prof MD, Principal Investigator — University Clinic of Hamburg-Eppendorf; 20246 Hamburg / Germany
Locations (4):
- Innsbruck, Austria
- Hamburg, Berlin, Heidelberg, Köln, Halle, Germany
- Terrassa, Spain
- Nottingham, United Kingdom

REFERENCES:
- [Background] Heiss MM, Strohlein MA, Jager M, Kimmig R, Burges A, Schoberth A, Jauch KW, Schildberg FW, Lindhofer H. Immunotherapy of malignant ascites with trifunctional antibodies. Int J Cancer. 2005 Nov 10;117(3):435-43. doi: 10.1002/ijc.21165. PMID 15906359
- [Background] Ruf P, Lindhofer H. Induction of a long-lasting antitumor immunity by a trifunctional bispecific antibody. Blood. 2001 Oct 15;98(8):2526-34. doi: 10.1182/blood.v98.8.2526. PMID 11588051
- [Background] Riesenberg R, Buchner A, Pohla H, Lindhofer H. Lysis of prostate carcinoma cells by trifunctional bispecific antibodies (alpha EpCAM x alpha CD3). J Histochem Cytochem. 2001 Jul;49(7):911-7. doi: 10.1177/002215540104900711. PMID 11410615
- [Background] Zeidler R, Mysliwietz J, Csanady M, Walz A, Ziegler I, Schmitt B, Wollenberg B, Lindhofer H. The Fc-region of a new class of intact bispecific antibody mediates activation of accessory cells and NK cells and induces direct phagocytosis of tumour cells. Br J Cancer. 2000 Jul;83(2):261-6. doi: 10.1054/bjoc.2000.1237. PMID 10901380
- [Background] Zeidler R, Reisbach G, Wollenberg B, Lang S, Chaubal S, Schmitt B, Lindhofer H. Simultaneous activation of T cells and accessory cells by a new class of intact bispecific antibody results in efficient tumor cell killing. J Immunol. 1999 Aug 1;163(3):1246-52. PMID 10415020